CLINICAL TRIAL: NCT00921037
Title: First Clinical Study of Erbium-YAG Laser Vaporisation of Cutaneous Neurofibromas
Brief Title: First Clinical Study of Erbium - Yttrium Aluminium Garnet (YAG) Laser Vaporization of Cutaneous Neurofibromas
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Wolfgang Happak, Prof. MD, Division of Plastic and Reconstructive Surgery, Surgical Clinic, Medical University of Vienna, Austria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK Nr: 128/2006
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2009-06

CONDITIONS: Cutaneous Neurofibromas
Keywords: Neurofibromatosis Type 1; Morbus Recklinghausen; cutaneous neurofibromas; Erbium-YAG-Laser; Vaporisation; Thermal Necrosis
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erbium YAG Laser (Experimental): Patients with Neurofibromatosis Type 1 (Recklinghausen)
  Interventions: Procedure: Erbium-YAG laser vaporization

INTERVENTIONS:
Procedure: Erbium-YAG laser vaporization — spot size 2-5 mm diameter, applying about 1,2 -2 J at a frequency of 6-12 Hz

SUMMARY:
The purpose of this study is to determine whether multiple cutaneous neurofibromas in patients with neurofibromatosis type 1 can be removed with an erbium-YAG-laser.

DETAILED DESCRIPTION:
With a prevalence of 1 in 3-5000 births, neurofibromatosis Type I is one of the most common genetic defects. The mode of inheritance is autosomal dominant and affects a gene (NF1), which is responsible for the production of the tumor suppressor protein neurofibromin. The consequence is an uninhibited expansion of neural tissue which leads amongst others to cosmetic disfigurement of the patients. In comparison to the plexiform neurofibromas the cutaneous tumors do not undergo malignant transformation.

Excision and CO2 laser vaporisation were established as standard treatment but cause unattractive scars.

In one operation more than 500 neurofibromas can be removed with an Erbium: YAG laser (2940 nm). The tumors are dissected by shooting holes into the skin and vaporising the neurofibromas in-between or underneath. Specimen are harvested after Er: YAG-, CO2 - and electrosurgical treatment to evaluate the difference of thermal necrosis histologically and photographs are taken to assess the cosmetic results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple cutaneous neurofibromas with the request for tumor removal

Exclusion Criteria:

* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-04; Primary Completion 2012-01 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to enhance the quality of life (measured by the Nottingham Health Profile the Rosenberg's Self-Esteem Scale and the SF-36 health survey) of patients suffering from disfigurement due to thousands of cutaneous neurofibromas. | 6 months
  The standardized questionnaires are done before and 6 month after the operation in which the tight tumor cluster are phased down and thereby an almost normal skin appearance is achieved.

SECONDARY OUTCOMES:
With this new method we want to decrease the painfulness, accelerated the time till wound healing as well as reduce the stay in hospital and the incidence of side effects. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Happak, Prof. MD, Principal Investigator — Division of Plastic and Reconstructive Surgery, Surgical Clinic, Medical University of Vienna, Austria
Locations (1):
- Division of Plastic and Reconstructive Surgery, Surgical Clinic, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Algermissen B, Müller U, Katalinic D, Berlien HP. Laserbehandlung von kutanen Neurofibromen. journalmed. 12; 2001.
- [Background] Becker DW Jr. Use of the carbon dioxide laser in treating multiple cutaneous neurofibromas. Ann Plast Surg. 1991 Jun;26(6):582-6. doi: 10.1097/00000637-199106000-00016. PMID 1909107
- [Background] Kardorff B. Neurofibromatose Typ I (Morbus Recklinghausen): Kombinierte Erbium.Yag-Laser- und Exzisionstherapie von kutanen Neurofibromen. Derm 1998; 4:404-406
- [Background] Moreno JC, Mathoret C, Lantieri L, Zeller J, Revuz J, Wolkenstein P. Carbon dioxide laser for removal of multiple cutaneous neurofibromas. Br J Dermatol. 2001 May;144(5):1096-8. doi: 10.1046/j.1365-2133.2001.04214.x. No abstract available. PMID 11359412
- [Background] Ostertag JU, Theunissen CC, Neumann HA. Hypertrophic scars after therapy with CO2 laser for treatment of multiple cutaneous neurofibromas. Dermatol Surg. 2002 Mar;28(3):296-8. doi: 10.1046/j.1524-4725.2002.01145.x. PMID 11896787
- [Background] Querings K, Fuchs D, Kung EE, Hafner J. [CO2-laser therapy of stigmatizing cutaneous lesions in tuberous sclerosis (Bourneville-Pringle) and in neurofibromatosis 1 (von Recklinghausen)]. Schweiz Med Wochenschr. 2000 Nov 11;130(45):1738-43. German. PMID 11109606
- [Background] Roenigk RK, Ratz JL. CO2 laser treatment of cutaneous neurofibromas. J Dermatol Surg Oncol. 1987 Feb;13(2):187-90. doi: 10.1111/j.1524-4725.1987.tb00517.x. PMID 3100595